CLINICAL TRIAL: NCT00848497
Title: Efficacy of Testosterone Replacement Therapy in Penile Rehabilitation Following Radical Prostatectomy (#: 04-07-30-01)
Brief Title: Testosterone for Penile Rehabilitation After Radical Prostatectomy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of volunteers who would consent to participate and lack of funding
Sponsor: Mohit Khera (Other)
Responsible Party: Sponsor-Investigator, Mohit Khera, Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-21148
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Hypogonadism; Erectile Dysfunction
Keywords: hormone replacement therapy; radical prostatectomy; erectile dysfunctions; scheduled for removal of prostate gland
MeSH Terms: conditions — Hypogonadism; Erectile Dysfunction | interventions — Testosterone; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testim® + Viagra® (Active Comparator): Testim® gel (50 mg of testosterone) once daily + Viagra® 25 mg tablet every night
  Interventions: Drug: Testim®; Drug: Viagra®
- Placebo Testim® + Viagra® (Placebo Comparator): Placebo Testim® gel once daily + Viagra® 25 mg tablet every night
  Interventions: Other: Placebo Testim®; Drug: Viagra®

INTERVENTIONS:
Drug: Testim® — Testim® 5 g of gel (one tube) containing 50 mg of testosterone once daily. This was the dose given to the patient which he started.
  Other Names: Testim® is the brand name for testosterone gel.
  Arms: Testim® + Viagra®
Other: Placebo Testim® — Placebo Testim® 5 g of gel (one tube)
  Other Names: Placebo Testim
  Arms: Placebo Testim® + Viagra®
Drug: Viagra® — Viagra 25mg was the dose given to the patient which he started.
  Other Names: Viagra® is the brand name for sildenafil citrate.; Viagra® 25 mg tablet daily at night

SUMMARY:
The purpose of this study is to determine the effectiveness of testosterone replacement therapy (TRT) in men following surgery to remove the prostate in improving erectile function. Subjects will be randomized (like flipping a coin) to one of two groups. One group will receive Testim® (testosterone gel) 5 g per day plus Viagra 25 mg every night and the other will receive Placebo-Testim® 5 g per day plus Viagra 25 mg every night.

Subjects will begin drug treatment 3 months after the initial screening visit and will take study drug for 3 months only. Participation will end at the end of the 6-month visit.

DETAILED DESCRIPTION:
There was only one patient who began treatment with the study drug. After blind was broken, it was noted that he received placebo Testim and Viagra.

ELIGIBILITY:
Inclusion Criteria:

* Males, 18 years of age or older, with low testosterone levels.
* Must have undergone a bilateral nerve sparing radical prostatectomy.
* Nadir PSA (Prostate-Specific Antigen) values should be less than 0.01 ng/ml on two consecutive occasions separated by 4 weeks at the start of treatment.
* Must give informed consent.
* Must be willing to complete follow-up visits.

Exclusion Criteria:

* Testosterone level greater than 300 ng/ dl
* Hemoglobin level greater than 18 ng/dl.
* Positive surgical margins or evidence of residual prostate cancer after surgery.
* Clinically suspected advanced disease or actual evidence of metastatic prostate cancer.
* Primary Gleason Grade greater than 3 or secondary Gleason Grade greater than 4 in the final pathologic specimen will be excluded.
* Taking nitrates or with contraindications to the use of Viagra or androgen therapy will be excluded.
* Known hypersensitivity to any component of the tablet will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Khera, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Khera M, Grober ED, Najari B, Colen JS, Mohamed O, Lamb DJ, Lipshultz LI. Testosterone replacement therapy following radical prostatectomy. J Sex Med. 2009 Apr;6(4):1165-1170. doi: 10.1111/j.1743-6109.2009.01161.x. Epub 2009 Jan 22. PMID 19207277
- [Background] Khera M, Lipshultz LI. The role of testosterone replacement therapy following radical prostatectomy. Urol Clin North Am. 2007 Nov;34(4):549-53, vi. doi: 10.1016/j.ucl.2007.08.007. PMID 17983894
- [Background] Khera M. Androgens and erectile function: a case for early androgen use in postprostatectomy hypogonadal men. J Sex Med. 2009 Mar;6 Suppl 3:234-8. doi: 10.1111/j.1743-6109.2008.01159.x. Epub 2009 Jan 21. PMID 19207279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was approved for enrollment on 11/28/2007 and was closed on 1/25/13. Participants were consented in the Baylor Urology clinic setting.
Groups:
- Testim + Viagra: Testim® gel (50 mg of testosterone)once daily + Viagra® 25 mg tablet every night
- Placebo Testim + Viagra: Placebo Testim® gel (50 mg of testosterone) once daily + Viagra® 25 mg tablet every night
Period: Overall Study
Arm/Group | Testim + Viagra | Placebo Testim + Viagra
Started | 2 | 1 (Completed Visit 4)
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Screen failure | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Arm 1 = 2 Arm 2 = 1
Groups:
- Arm 1: Testim® gel (50 mg of testosterone)once daily + Viagra® 25 mg tablet every night
- Arm 2: Placebo Testim® gel (50 mg of testosterone) once daily + Viagra® 25 mg tablet every night
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (4) | 59 (0) | 56 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in SHIM (Sexual Health Inventory for Males) Score at 6 Months After Initial Screening Visit.
Description: SHIM range is 0-25. 0= no sexual activity;1-7 severe ED; 8-11 Moderate ED; 12-16 Mild to Moderate ED; 17-21 Mild ED
Time Frame: Baseline and 6 months
Population: Baseline = 0 5 months = 0
Measure: Number; unit: units on a scale
Groups:
- Testim + Viagra: Testim® gel (50 mg of testosterone)once daily + Viagra® 25 mg tablet every night
  SHIM at Baseline = N/A SHIM at 5 months = N/A
- Placebo Testim + Viagra: Placebo Testim® gel (50 mg of testosterone) once daily + Viagra® 25 mg tablet every night
  SHIM at Baseline = 0 SHIM at 5 months = 0
Arm/Group | Testim + Viagra | Placebo Testim + Viagra
Number analyzed (Participants) | 0 | 1
units on a scale |  | 0

2. Secondary Outcome: Change in the IIEF (International Index of Erectile Function) Score 6 Months After the Initial Screening Visit.
Description: There are 15 questions, each divided into 5 domains. Maximum score is 75 = best function, and minimum is 5 = worst function
Time Frame: Baseline and 6 months
Population: Baseline = 5 5 months = 6
Measure: Number; unit: units on a scale
Arm/Group | Testim + Viagra | Placebo Testim + Viagra
Number analyzed (Participants) | 0 | 1
units on a scale |  | 1

3. Secondary Outcome: Change in the ADAM (Androgen Deficiency in the Aging Male)Score 6 Months After the Initial Screening Visit.
Description: ADAM scores of one evaluated patient. ADAM is 10 questions ("yes" or "no" answers) and if you answer yes to question 1 or 7 or "yes" to any 3 questions you are said to test "positive" to the ADAM questionnaire.
Time Frame: Baseline and 6 months
Population: Baseline = Positive 5 months = Positive
Measure: Number; unit: number of yes answers
Arm/Group | Testim + Viagra | Placebo Testim + Viagra
Number analyzed (Participants) | 0 | 1
number of yes answers |  | 1

4. Secondary Outcome: Change in the EPIC (Expanded Prostate Cancer Index Composite) Score 6 Months After the Initial Screening Visit.
Description: EPIC is scored from 0 -100,lower EPIC score= worse, higher EPIC score= better
Time Frame: Basline and 6 months
Population: Baseline = 98
  5 months = 87
Measure: Number; unit: units on a scale
Arm/Group | Testim + Viagra | Placebo Testim + Viagra
Number analyzed (Participants) | 0 | 1
units on a scale |  | -11

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
The subject that completed the study reported no adverse reactions or events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No